CLINICAL TRIAL: NCT06209320
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Phase III Clinical Study of the Efficacy and Safety of Two Low-concentration Atropine Sulfate Eye Drops in Slowing the Progression of Myopia in Children
Brief Title: A Study of the Efficacy and Safety of Two Low-concentration Atropine Sulfate Eye Drops
Acronym: China-CHAMP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZKO-ATP-202105-China-CHAMP
Record Dates: First submitted 2024-01-06; First posted 2024-01-17 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental group 1 (Active Comparator): Lower dose atropine sulfate eye drops
  Interventions: Drug: Lower dose atropine sulfate eye drops
- Experimental group 2 (Active Comparator): Low dose atropine sulfate eye drops
  Interventions: Drug: Low dose atropine sulfate eye drops
- control group (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Lower dose atropine sulfate eye drops — administer to eyes
  Other Names: Lower dose atropine sulfate
  Arms: Experimental group 1
Drug: Low dose atropine sulfate eye drops — administer to eyes
  Other Names: Low dose atropine sulfate
  Arms: Experimental group 2
Drug: placebo — administer to eyes
  Other Names: Vehicle
  Arms: control group

SUMMARY:
A randomized, double-blind, placebo-controlled, multicenter, phase III clinical study of the efficacy and safety of two low-concentration atropine sulfate eye drops in slowing the progression of myopia in children

DETAILED DESCRIPTION:
Primary objective is to evaluate the efficacy and safety of atropine sulfate eye drops versus placebo for 12 months in slowing the progression of myopia in children.

The study was designed to enroll approximately 777 subjects. Eligible subjects were randomly assigned to the placebo control group, Lower dose atropine group and Lower dose atropine group. Subjects received the study medication in both eyes, 1 drop each time, once every night at bedtime.

Statistical analyses were performed with the use of SAS software, version 9.4, without any specific description. All statistical tests were two-sided at a 0.05 level.

ELIGIBILITY:
Inclusion Criteria:

1. Child (female or male) aged 6 to 12 years.
2. Myopia (SER of at least -0.50 D and no more myopic than -6.00 D) in each eye as measuredby cycloplegic autorefraction.
3. If present, astigmatism of ≤1.50 D in each eye as measured by cycloplegic autorefraction.
4. Anisometropia SER of < 1.50 D as measured by cycloplegic autorefraction.

Exclusion Criteria:

1. Have used other myopia control methods other than those used in this study, such as instruments (orthokeratology lenses, multifocal glasses, progressive glasses), drugs (atropine, etc.); Only single vision glasses are allowed for myopia correction;
2. Have used myopic control methods such as traditional Chinese medicine, auricular acupuncture, massage, and reverse beat within 30 days before screening;
3. Use of any local or systemic antimuscarinic/anticholinergic medication (e.g., atropine, scopolamine, tropicamide, phenamine, diphenhydramine, oxytropine, tricyclic antidepressant, etc.) within 21 days before screening; Allowing for tests such as cycloplegic optometry;

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 777 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Cycloplegic Autorefraction(SER) | 24 months
  Between-group difference in the mean change from baseline in SER at visit M24

SECONDARY OUTCOMES:
Axial Length | 24 months
  Between-group difference in the mean change from baseline in axial length at visit M24

OTHER OUTCOMES:
Relationship between age and slow myopia progression | 24 months
  Relationship between age and slow in myopia progression (SER change from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Ningli Wang, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China